CLINICAL TRIAL: NCT01915186
Title: A Randomized Controlled Trial on the Effect of Dehydroepiandrosterone (DHEA) Supplementation on Ovarian Reserve Markers, Response to a Standard Low Dose FSH Stimulation and IVF Cycle Outcomes in Patients With Normal and Poor Ovarian Reserve
Brief Title: Use of Dehydroepiandrosterone (DHEA) in Women With Normal and Poor Ovarian Reserve Undergoing IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yeung Wing Yee Tracy, Associate Consultant, The University of Hong Kong
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: TY-02
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Female Infertility Due to Diminished Ovarian Reserve
Keywords: DHEA; Poor ovarian reserve; Normal ovarian reserve; In vitro fertilization treatment; Ovarian response; Pregnancy outcomes
MeSH Terms: interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dihydroepiandrosterone (DHEA) (Experimental): DHEA 25mg 3 times a day for 12 weeks
  Interventions: Dietary Supplement: Dihydroepiandrosterone (DHEA)
- Placebo (Placebo Comparator): Matched placebo capsules are given 3 times a day for 12 weeks

INTERVENTIONS:
Dietary Supplement: Dihydroepiandrosterone (DHEA) — DHEA capsules are given at 25mg 3 times a day for 12 weeks
  Other Names: DHEA (GNC)
  Arms: Dihydroepiandrosterone (DHEA)

SUMMARY:
The aim of the study is to evaluate the effect of DHEA supplement on ovarian reserve markers, ovarian response to gonadotrophins and cycle outcomes in patients with normal and poor ovarian reserve.

Study Hypotheses:

1. DHEA supplementation would improve markers of ovarian reserve and ovarian response to low dose FSH stimulation in both normal and poor responders
2. DHEA supplementation would improve IVF cycle outcomes

DETAILED DESCRIPTION:
Consecutive patients attending subfertility clinic at the Department of Obstetrics and Gynaecology, Queen Mary Hospital who are scheduled for in-vitro fertilization (IVF) treatment will be recruited and written consent will be obtained.

Baseline assessment will be performed at early follicular phase (Day 2 or 3) with hormonal tests and ultrasound.

Subjects will be divided into two groups, the normal ovarian reserve group and the poor ovarian reserve group according to AFC. Poor ovarian reserve is defined as an AFC of less than 5, while normal ovarian reserve is defined as an AFC of 5 to 15 based on a previous study showing AFC being a good predictor of ovarian response (Tomas 1997). Subjects with normal ovarian reserve will be further subdivided into <35 and >/=35 years old while subjects with poor ovarian reserve will be further subdivided into first or subsequent cycles of IVF for subgroup analysis.

Subjects in both the normal and poor ovarian reserve group will be randomized according to a computer-generated randomization list in sealed envelopes to receive either DHEA at 25mg three times a day or placebo throughout the study period.

Any changes in hormonal profile and ovarian reserve will be assessed by the above-mentioned blood tests and pelvic ultrasound scans which will be repeated at early follicle phase (Day 2 or 3) in the two subsequent cycles.

After two months of DHEA/placebo treatment, the subjects will then be given a standard low dose ovarian stimulation with 75 IU intramuscular human menopausal gonadotrophin (HMG, Menogon®, Ferring Pharmaceuticals) daily for 7 days. Blood tests and pelvic ultrasound scan will be repeated after 7 days of stimulation (ie. on day 10 or 11).

Hormonal profile and ovarian reserve will be repeated in follicular phase (D2 or 3) in the subsequent cycle, where all patients will then be offered a cycle of IVF treatment using antagonist protocol based on our standard departmental regimen. Cycle characteristic and pregnancy outcomes will be compared.

Analysis of ovarian reserve markers, ovarian response and IVF outcomes would be performed.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for IVF treatment according to our standard department protocol
* Age < 40
* Regular menstrual cycles (21-35 days with </= 4 days inter-cycle variation)
* AFC not more than 15

Exclusion Criteria:

* Previous chemotherapy or pelvic irradiation
* Polycystic ovarian syndrome or polycystic ovaries
* On hormonal supplementation for any indication at the time of recruitment (e.g. estrogen, testosterone or DHEA)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Antral follicle count | after 12 weeks of DHEA
  Compare the changes in antral follicle count after 12 weeks of DHEA supplementation prior to IVF treatment between the treatment and placebo groups

SECONDARY OUTCOMES:
Change in Follicular stimulating hormone (FSH) and anti-Mullerian Hormone (AMH) following DHEA supplementation; post stimulation estradiol level and number of follicles > 10mm, IVF outcomes, hormonal profile of follicular fluid | after 12 weeks of DHEA
  Comparison on the ovarian reserve markers, response to low dose ovarian stimulation and IVF treatment outcomes between treatment and control groups

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Gleicher N, Barad DH. Dehydroepiandrosterone (DHEA) supplementation in diminished ovarian reserve (DOR). Reprod Biol Endocrinol. 2011 May 17;9:67. doi: 10.1186/1477-7827-9-67. PMID 21586137
- [Derived] Yeung TW, Chai J, Li RH, Lee VC, Ho PC, Ng EH. A randomized, controlled, pilot trial on the effect of dehydroepiandrosterone on ovarian response markers, ovarian response, and in vitro fertilization outcomes in poor responders. Fertil Steril. 2014 Jul;102(1):108-115.e1. doi: 10.1016/j.fertnstert.2014.03.044. Epub 2014 May 3. PMID 24796766